CLINICAL TRIAL: NCT00664651
Title: Capsular Changes in Joint Contractures Post-Knee Arthroplasty:A Case-Control Study
Brief Title: Joint Stiffness Following Knee Replacement Surgery
Status: Withdrawn | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Guy Trudel, Researcher, Ottawa Hospital Research Institute
Other Study IDs: 2006541
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Joint Contracture
Keywords: joint contracture; total knee arthroplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Our primary research question is to find out whether there is a genetic component to the development of joint contractures following knee surgery, through the application of lab techniques.

DETAILED DESCRIPTION:
After total knee replacement surgery, some people develop joint stiffness, which is also called a joint contracture. Contractures cause the envelope of the knee (called the capsule) to stiffen and become rigid so the patient can no longer move their knee the way they used to. After stretching and other exercises, only a surgery can try and divide or remove the contracture. The main purpose of this research is to study the cause of the contracture and specifically if certain people are predisposed to contractures.

ELIGIBILITY:
Inclusion Criteria:

-knee contractures post arthroplasty scheduled for arthrotomy with debridement of capsular tissue Controls will be patients scheduled for arthrotomy with debridement of capsular tissue for the other reasons(primary knee arthroplasty, ORIF of the knee secondary to trauma, ACL repair, amputation, elective joint arthroplasty with capsuloplasty etc.)

Exclusion:

* transmissible disease (HIV, Hep B,C)
* confirmed or suspected neoplasia
* suspected infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: joint contractures following knee surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Gene expression | Dec 2015

CONTACTS AND LOCATIONS:
Overall Officials: Guy Trudel, MD,MSc,FRCPC, Principal Investigator — OHRI / The Ottawa Hospital
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada